CLINICAL TRIAL: NCT04691232
Title: Phase I, Open-label, Fast-track Dose-escalation Clinical Trial Exploring the Safety and the Tolerability of Autologous ex Vivo Expanded Regulatory T Cells in Adults With Ulcerative Colitis
Brief Title: Autologous Ex Vivo Expanded Regulatory T Cells in Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ER-TREG 01
Record Dates: First submitted 2020-12-07; First posted 2020-12-31 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2022-01

CONDITIONS: Ulcerative Colitis; Autoimmune Diseases
Keywords: Ulcerative colitis; Regulatory T cells; Adoptive cell therapy
MeSH Terms: conditions — Colitis, Ulcerative; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regulatory T cells (Experimental): Intravenous infusion of a single dose of 0.5x10e6, 1x10e6, 2x10e6, 5x10e6 or 10x10e6 Treg/kg body weight
  Interventions: Biological: Regulatory T cells

INTERVENTIONS:
Biological: Regulatory T cells — Autologous, ex vivo expanded, regulatory T cells

SUMMARY:
Together with Crohn's disease (CD), ulcerative colitis (UC) is one of the major forms of inflammatory bowel diseases (IBD).Currently, no curative therapy is available, since the pathophysiology of this disease is incompletely understood (1-3) and clinical practice demonstrates that current therapies induce remission in subgroups of patients only. Scientific evidence suggests that colitogenic immune responses can be controlled by increasing the number of circulating regulatory T cells (Treg) (4). The production of large numbers of autologous Treg is possible by isolation of CD25+ cells from the whole blood of a patient and subsequent ex vivo expansion in the presence of the immunomodulatory drug rapamycin, Interleukin-2 (IL-2) and CD3/CD28 expander beads (5).

ER-TREG 01 is a single-center, open-label, fast-track phase I dose-escalation study designed to assess the safety profile and maximal tolerated dose (MTD) of a single infusion of ex vivo expanded autologous Treg in patients with active ulcerative colitis.

DETAILED DESCRIPTION:
While the primary cause of inflammatory bowel disease (IBD) development remains unknown, it is widely accepted that the initial events culminate in persistent immune responses with infiltration of immune cells and tissue destruction in the gut. Immune cell populations present within the inflamed bowel wall of IBD patients have been extensively characterized and studied (1;6). Studies focusing on T cells have demonstrated that the mucosa of Crohn's disease (CD) patients is dominated by Th1 cells, while in patients with ulcerative colitis (UC) T helper cells with an atypical Th2 profile, which excessively produce IL-5 and IL-13 but not IL-4, are abundant (7). Furthermore, Th17 cells can be identified in the inflamed lamina propria and these cells are thought to play an important role in the pathophysiology of IBD, although the pathogenic mechanisms of these cells are not yet fully understood (8;9). Treg are also present within the lamina propria and these cells control the effector T cell populations mentioned above. They can be generated through the interaction of local T cells with CD103 expressing dendritic cells and intestinal epithelial cells, respectively (10;11). Moreover, the expression of integrins on the Treg surface (e.g. α4β7) facilitates mucosal migration through their interaction with specific ligands (e.g. MAdCAM1). As such, homing and local expansion of Treg cells create a local Treg pool that is essential for self-tolerance and the support of gut homeostasis (12). In addition, Treg cells are shown to suppress proinflammatory intestinal immune responses in colitis and colitis-associated cancer (13-16) and they are thought to augment intestinal Th17 responses (17). As previous studies have demonstrated insufficient expansion of mucosal Treg cells in IBD patients in comparison to the massive local expansion of effector T cells, it is likely that the relatively low number of Treg cells in IBD patients explains why these cells fail to control excessive immune responses (18).

Experimental colitis studies in mice have demonstrated that colitogenic immune responses can be controlled by increasing the number of mucosal Treg cells and highlight the potential of Treg-based cell therapy in IBD (19). Specifically, co-transfer of naïve CD4+ T cells with Treg both prevents chronic colitis and ameliorates established colitis in severe combined immunodeficiency (SCID) mice (20). Moreover, CD4+ T cells expanded ex vivo in the presence of rapamycin prevent the development of colitis in a naïve CD4+ T cell model in SCID mice. Importantly, the systemic administration of rapamycin alone only partially prevented the development of colonic Inflammation (20). In addition, the adoptive transfer of nTreg cells as well as the adoptive transfer of ex vivo transforming growth factor (TGF)-β-induced Treg (iTreg) suppressed colitis activity in vivo in mouse models (13;15;21). Collectively, these data suggest that Treg cells could be used for therapy of intestinal inflammation in IBD (22).

To allow an adoptive transfer of large numbers of Treg, CD25+ Treg cells are isolated from an autologous leukapheresis product and in vitro expanded during 21 days in the presence of the additives Interleukin-2 (IL-2), rapamycin and anti-CD3/anti-CD28 expander beads. After 21 days of expansion, anti-CD3/anti-CD28 expander beads are removed from the Treg drug product. Next, Treg are frozen in aliquots of 10 Million Treg/mL until further use (5).

Twelve patients, including 10% patient loss, resulting in at least ten treated and fully evaluable patients, will be enrolled in this single-center, open-label, fast-track dose-escalation study. Autologous ex vivo expanded CD4+CD25+CD127-/lo Treg cells will be adoptively transferred in patients with ulcerative colitis with active disease or stable disease under the allowed concomintant therapy at the time of enrollment. The maximal tolerated dose (MTD) is defined as the dose that does not produce more than one dose-limiting toxicity (DLT) among a total of four treated patients at the particular dose level.

The first enrolled patient will receive the initial starting dose of 0.5 x10e6 Treg/kg bodyweight. Adoptive transfer is escalated to the next dose level (1 x 10e6 Treg/kg, 2 x 10e6 Treg/kg, 5 x 10e6/Treg/kg and 10 x 10e6 Treg/kg bodyweight), in a next patient, if no DLT occurs. Consecutive patients will be treated at least four weeks apart to monitor acute severe adverse advents. If a DLT is noted, three additional patients will receive the same dose level. Dose-escalation continues until at least two patients among a cohort of four patients experience a DLT. If two patients among a cohort of four patients experience a DLT, dose de-escalation to the highest previously tolerated dose-level will follow. Three additional patients will receive the highest previously tolerated dose. If a DLT is noted in at least two patients at the tested dose-level, dose de-escalation will continue until less than two patients have experienced a DLT. After successful enrollment at the highest dose-level, five additional patients will be enrolled at the highest dose level to extend safety assessment. If no DLTs or less than two DLTs are experienced at all dose-levels tested, the MTD is not reached. In this case, a maximal administered dose (MAD) is defined.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an established diagnosis of UC, with minimum time from diagnosis of ≥3 months
* Patients must be either in remission under the allowed concomitant therapy or must have received all the beneficial pharmacological treatment lines before enrollment and have moderate to severe disease activity (disease should extend 15 cm or more above the anal verge) determined by a modified Mayo score (excluding the friability at grade 1 for the endoscopic sub score) of 6 to 12 with an endoscopic subscore ≥ 2 and no other individual subscore < 1.
* Patients must have a WHO performance status of 0, 1 or 2 and must be in stable medical condition.
* Patients must be between 18 and 75 years old and must be able and willing to give informed consent.
* Women of child-bearing age must have a negative pregnancy test at enrollment in the study, must be willing to undergo monthly pregnancy tests until at least 3 months after adoptive Treg transfer and must oblige to use effective contraception until at least 3 months after adoptive Treg transfer. A highly effective method of birth control is defined as one that results in a low failure rate (ie, less than 1 percent per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner. For subjects using a hormonal contraceptive method, information regarding the product under evaluation and its potential effect on the contraceptive should be addressed.
* Male study patients, who are partners of women of child-bearing age must be willing to use effective contraception until at least 3 months after adoptive Treg transfer. A highly effective method of birth control is defined as one that results in a low failure rate (ie, less than 1 percent per year) when used consistently and correctly, such as sexual abstinence, or a vasectomy. The solely use of condoms is not considered as an effective method of birth control. Therefore, partners of child-bearing age from male study patients should be willing to use implants, injectables, combined oral contraceptives or intrauterine devices (IUDs) a highly effective method of birth control. Information regarding the product under evaluation and its potential effect on the contraceptive should be addressed.
* Patients must be willing to undergo a leukapheresis.
* Patients must be willing to get hospitalized for at least 24 hours following adoptive Treg transfer, and to cooperate for the whole period of the trial.
* Accomplishment of a washout phase for biological therapy of at least 8 weeks or no detectable serum trough levels prior to screening in case of a washout phase less than 8 weeks.
* Concomitant therapy with oral corticosteroids (prednisone or equivalent up to 20 mg/day, stable for 2 weeks at inclusion), budesonide (9 mg/day, stable for 8 weeks at inclusion), 5-ASA (stable for 2 weeks at inclusion) and azathioprine (stable for 8 weeks, initiated at least 3 months ago) is permitted. Concomitant oral corticosteroids can be reduced at the investigator's discretion from visit 5 onwards (e.g. 5 mg reduction per week).≤

Exclusion Criteria:

* Any of the above mentioned inclusion criteria are not met.
* Impaired hematological function (on repeated testing) as indicated by Leukocyte Count ≤ 2,500 /mm3, or Neutrophils ≤ 1,000 / mm3, or Lymphocytes ≤ 700 / mm3, or Platelets ≤ 75,000 / mm3, or Hemoglobin ≤ 9 g / dl22
* Impaired hepatic or renal function as indicated by Serum creatinine ≥ 2.5 mg/100 ml, or Serum Bilirubin ≥ 2.0 mg/100 ml
* Any other major serious illness [e.g. active systemic infections, immunodeficiency disease, clinically significant heart disease, respiratory disease, bleeding disorders, etc.] or a contraindication to leukapheresis.
* Evidence for HIV-1, HIV -2, HTLV-1, TPHA, HBV, or HCV infection.
* Patients who have spent a cumulative period of 1 year or more in the UK between the beginning of 1980 and the end of 1996
* Patients who have a family history, which places them at risk of developing Creutzfeldt-Jacob disease
* Patients who have received a corneal or dura mater graft, or who have been treated in the past with medicines made from human pituitary glands
* Other active autoimmune diseases (such as but not limited to Lupus erythematosus, autoimmune thyroiditis or uveitis, multiple sclerosis).
* Previous splenectomy or radiation therapy to the spleen.
* Patients with organ allografts.
* Patients with celiac disease.
* Concomitant treatment with chemotherapy, immunotherapy, any investigational drug and paramedical substances.
* Existence or prior history of a malignant neoplasm.
* Organic brain syndrome or significant psychiatric abnormality which would preclude participation in the full protocol and follow up.
* Positive pregnancy test / Pregnancy or lactation. If pregnancy occurs during the course of the trial to female patients, the patient has to be excluded (not valid for partners of male patients treated).
* Known hypersensitivities to human serum albumin and/or DMSO

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Dose-finding | Visit 5 (4 weeks after adoptive Treg transfer)
  To define the maximum tolerable dose (MTD) of one single infusion of autologous ex vivo expanded regulatory T cells in patients with ulcerative colitis

SECONDARY OUTCOMES:
Assessment of safety of one single Infusion of regulatory T cells | Visit 5 (4 weeks after adoptive Treg transfer)
  To define the number of patients with treatment-related adverse events as assessed by CTCAE v. 5.0
Assessment of inflammation in the gut | Visit 5 (4 weeks after adoptive Treg transfer)
  To define the impact on the course of UC as defined by an increase in the Mayo Clinic score of at least 3 points and an increase of at least 30% from baseline, with an accompanying increase in rectal bleeding subscore of at least 1 point.
Assessment of quality of life | Visit 5 (4 weeks after adoptive Treg transfer)
  To define changes in disease activity score calculated by the evaluation of the Quality of Life Inflammatory Bowel Disease Questionnaire (IBDQ)
Assessment of Treg function in peripheral blood | Visit 5 (4 weeks after adoptive Treg transfer)
  To define changes in Treg frequency in peripheral blood
Assessment of Treg function in the gut | Visit 5 (4 weeks after adoptive Treg transfer)
  To define changes in effector T cell and Treg frequencies in the gut

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Markus Neurath, MD, Principal Investigator — University of Erlangen-Nürnberg Medical School
Locations (1):
- University of Erlangen-Nürnberg Medical School, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abraham C, Cho JH. Inflammatory bowel disease. N Engl J Med. 2009 Nov 19;361(21):2066-78. doi: 10.1056/NEJMra0804647. No abstract available. PMID 19923578
- [Background] Corridoni D, Arseneau KO, Cominelli F. Inflammatory bowel disease. Immunol Lett. 2014 Oct;161(2):231-5. doi: 10.1016/j.imlet.2014.04.004. Epub 2014 Jun 2. PMID 24938525
- [Background] Danese S, Fiocchi C. Ulcerative colitis. N Engl J Med. 2011 Nov 3;365(18):1713-25. doi: 10.1056/NEJMra1102942. No abstract available. PMID 22047562
- [Background] Mayne CG, Williams CB. Induced and natural regulatory T cells in the development of inflammatory bowel disease. Inflamm Bowel Dis. 2013 Jul;19(8):1772-88. doi: 10.1097/MIB.0b013e318281f5a3. PMID 23656897
- [Background] Wiesinger M, Stoica D, Roessner S, Lorenz C, Fischer A, Atreya R, Neufert CF, Atreya I, Scheffold A, Schuler-Thurner B, Neurath MF, Schuler G, Voskens CJ. Good Manufacturing Practice-Compliant Production and Lot-Release of Ex Vivo Expanded Regulatory T Cells As Basis for Treatment of Patients with Autoimmune and Inflammatory Disorders. Front Immunol. 2017 Oct 26;8:1371. doi: 10.3389/fimmu.2017.01371. eCollection 2017. PMID 29123521
- [Background] Geremia A, Biancheri P, Allan P, Corazza GR, Di Sabatino A. Innate and adaptive immunity in inflammatory bowel disease. Autoimmun Rev. 2014 Jan;13(1):3-10. doi: 10.1016/j.autrev.2013.06.004. Epub 2013 Jun 15. PMID 23774107
- [Background] Neurath MF. Cytokines in inflammatory bowel disease. Nat Rev Immunol. 2014 May;14(5):329-42. doi: 10.1038/nri3661. Epub 2014 Apr 22. PMID 24751956
- [Background] Iboshi Y, Nakamura K, Fukaura K, Iwasa T, Ogino H, Sumida Y, Ihara E, Akiho H, Harada N, Nakamuta M. Increased IL-17A/IL-17F expression ratio represents the key mucosal T helper/regulatory cell-related gene signature paralleling disease activity in ulcerative colitis. J Gastroenterol. 2017 Mar;52(3):315-326. doi: 10.1007/s00535-016-1221-1. Epub 2016 May 13. PMID 27178567
- [Background] Sujino T, Kanai T, Ono Y, Mikami Y, Hayashi A, Doi T, Matsuoka K, Hisamatsu T, Takaishi H, Ogata H, Yoshimura A, Littman DR, Hibi T. Regulatory T cells suppress development of colitis, blocking differentiation of T-helper 17 into alternative T-helper 1 cells. Gastroenterology. 2011 Sep;141(3):1014-23. doi: 10.1053/j.gastro.2011.05.052. Epub 2011 Jun 7. PMID 21699791
- [Background] Siddiqui KR, Powrie F. CD103+ GALT DCs promote Foxp3+ regulatory T cells. Mucosal Immunol. 2008 Nov;1 Suppl 1:S34-8. doi: 10.1038/mi.2008.43. PMID 19079226
- [Background] Westendorf AM, Fleissner D, Groebe L, Jung S, Gruber AD, Hansen W, Buer J. CD4+Foxp3+ regulatory T cell expansion induced by antigen-driven interaction with intestinal epithelial cells independent of local dendritic cells. Gut. 2009 Feb;58(2):211-9. doi: 10.1136/gut.2008.151720. Epub 2008 Oct 2. PMID 18832523
- [Background] Hadis U, Wahl B, Schulz O, Hardtke-Wolenski M, Schippers A, Wagner N, Muller W, Sparwasser T, Forster R, Pabst O. Intestinal tolerance requires gut homing and expansion of FoxP3+ regulatory T cells in the lamina propria. Immunity. 2011 Feb 25;34(2):237-46. doi: 10.1016/j.immuni.2011.01.016. Epub 2011 Feb 17. PMID 21333554
- [Background] Coombes JL, Maloy KJ. Control of intestinal homeostasis by regulatory T cells and dendritic cells. Semin Immunol. 2007 Apr;19(2):116-26. doi: 10.1016/j.smim.2007.01.001. Epub 2007 Feb 21. PMID 17320411
- [Background] Coombes JL, Siddiqui KR, Arancibia-Carcamo CV, Hall J, Sun CM, Belkaid Y, Powrie F. A functionally specialized population of mucosal CD103+ DCs induces Foxp3+ regulatory T cells via a TGF-beta and retinoic acid-dependent mechanism. J Exp Med. 2007 Aug 6;204(8):1757-64. doi: 10.1084/jem.20070590. Epub 2007 Jul 9. PMID 17620361
- [Background] Griseri T, Asquith M, Thompson C, Powrie F. OX40 is required for regulatory T cell-mediated control of colitis. J Exp Med. 2010 Apr 12;207(4):699-709. doi: 10.1084/jem.20091618. Epub 2010 Apr 5. PMID 20368580
- [Background] Pastille E, Bardini K, Fleissner D, Adamczyk A, Frede A, Wadwa M, von Smolinski D, Kasper S, Sparwasser T, Gruber AD, Schuler M, Sakaguchi S, Roers A, Muller W, Hansen W, Buer J, Westendorf AM. Transient ablation of regulatory T cells improves antitumor immunity in colitis-associated colon cancer. Cancer Res. 2014 Aug 15;74(16):4258-69. doi: 10.1158/0008-5472.CAN-13-3065. Epub 2014 Jun 6. PMID 24906621
- [Background] Wang Z, Friedrich C, Hagemann SC, Korte WH, Goharani N, Cording S, Eberl G, Sparwasser T, Lochner M. Regulatory T cells promote a protective Th17-associated immune response to intestinal bacterial infection with C. rodentium. Mucosal Immunol. 2014 Nov;7(6):1290-301. doi: 10.1038/mi.2014.17. Epub 2014 Mar 19. PMID 24646939
- [Background] Holmen N, Lundgren A, Lundin S, Bergin AM, Rudin A, Sjovall H, Ohman L. Functional CD4+CD25high regulatory T cells are enriched in the colonic mucosa of patients with active ulcerative colitis and increase with disease activity. Inflamm Bowel Dis. 2006 Jun;12(6):447-56. doi: 10.1097/00054725-200606000-00003. PMID 16775488
- [Background] Izcue A, Coombes JL, Powrie F. Regulatory T cells suppress systemic and mucosal immune activation to control intestinal inflammation. Immunol Rev. 2006 Aug;212:256-71. doi: 10.1111/j.0105-2896.2006.00423.x. PMID 16903919
- [Background] Ogino H, Nakamura K, Iwasa T, Ihara E, Akiho H, Motomura Y, Akahoshi K, Igarashi H, Kato M, Kotoh K, Ito T, Takayanagi R. Regulatory T cells expanded by rapamycin in vitro suppress colitis in an experimental mouse model. J Gastroenterol. 2012 Apr;47(4):366-76. doi: 10.1007/s00535-011-0502-y. Epub 2011 Dec 22. PMID 22189601
- [Background] Fantini MC, Becker C, Tubbe I, Nikolaev A, Lehr HA, Galle P, Neurath MF. Transforming growth factor beta induced FoxP3+ regulatory T cells suppress Th1 mediated experimental colitis. Gut. 2006 May;55(5):671-80. doi: 10.1136/gut.2005.072801. Epub 2005 Sep 14. PMID 16162681
- [Background] Salas A, Panes J. IBD. Regulatory T cells for treatment of Crohn's disease. Nat Rev Gastroenterol Hepatol. 2015 Jun;12(6):315-6. doi: 10.1038/nrgastro.2015.68. Epub 2015 Apr 21. PMID 25895817
- [Derived] Voskens C, Stoica D, Rosenberg M, Vitali F, Zundler S, Ganslmayer M, Knott H, Wiesinger M, Wunder J, Kummer M, Siegmund B, Schnoy E, Rath T, Hartmann A, Hackstein H, Schuler-Thurner B, Berking C, Schuler G, Atreya R, Neurath MF. Autologous regulatory T-cell transfer in refractory ulcerative colitis with concomitant primary sclerosing cholangitis. Gut. 2023 Jan;72(1):49-53. doi: 10.1136/gutjnl-2022-327075. Epub 2022 Apr 15. PMID 35428657
- [Derived] Voskens CJ, Stoica D, Roessner S, Vitali F, Zundler S, Rosenberg M, Wiesinger M, Wunder J, Siegmund B, Schuler-Thurner B, Schuler G, Berking C, Atreya R, Neurath MF. Safety and tolerability of a single infusion of autologous ex vivo expanded regulatory T cells in adults with ulcerative colitis (ER-TREG 01): protocol of a phase 1, open-label, fast-track dose-escalation clinical trial. BMJ Open. 2021 Dec 8;11(12):e049208. doi: 10.1136/bmjopen-2021-049208. PMID 34880013